CLINICAL TRIAL: NCT07000344
Title: A Multicenter, Open-Label, Prospective Cohort Study of Apatinib Plus Letrozole With or Without Fluzoparib as Second-Line Maintenance Therapy in ER-Positive, Platinum-Sensitive Recurrent Ovarian Cancer Following First-Line PARP Inhibitor Maintenance
Brief Title: A Study of Apatinib Combined With Letrozole With or Without Fluzoparib in Estrogen Receptor-Positive, Platinum-Sensitive Recurrent Ovarian Cancer Previously Treated With First-Line PARP Inhibitor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Fengzhi Feng, Chief Physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K7506
Record Dates: First submitted 2025-05-30; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; Platinum-Sensitive Recurrent; Maintenance Therapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (triple-drug group) (Experimental): Patients with advanced, estrogen receptor-positive, platinum-sensitive recurrent ovarian cancer who had previously received first-line poly (ADP-ribose) polymerase (PARP) inhibitor maintenance therapy.
  Interventions: Drug: Cohort 1 (triple-drug group)
- Cohort 2 (dual-drug group) (Experimental): Patients with advanced, estrogen receptor-positive, platinum-sensitive recurrent ovarian cancer who had previously received first-line poly (ADP-ribose) polymerase (PARP) inhibitor maintenance therapy.
  Interventions: Drug: Cohort 2 (dual-drug group)

INTERVENTIONS:
Drug: Cohort 1 (triple-drug group) — Apatinib: 250 mg orally once daily, with a 28-day treatment cycle. Fluzoparib: 100 mg orally twice daily, with a 4-week continuous treatment cycle.
  Letrozole: 2.5 mg orally once daily, with a 4-week continuous treatment cycle. Treatment continued until disease progression, intolerable toxicity, or other protocol-specified reasons occurred.
  Arms: Cohort 1 (triple-drug group)
Drug: Cohort 2 (dual-drug group) — Apatinib: 250 mg orally once daily, with a 28-day treatment cycle. Letrozole: 2.5 mg orally once daily, with a 4-week continuous treatment cycle. Treatment continued until disease progression, intolerable toxicity, or other protocol-specified reasons occurred.
  Arms: Cohort 2 (dual-drug group)

SUMMARY:
This multicenter, open-label, prospective cohort clinical study enrolled 70 patients with late-stage ER（+）platinum-sensitive recurrent ovarian cancer who had achieved CR/PR after first-line PARP inhibitor maintenance therapy. The study was divided into two cohorts, with 35 participants in each. Cohort 1 (triple-drug group) received the following treatments: Apatinib: 250 mg orally once daily, with a 28-day treatment cycle. Fluzoparib: 100 mg orally twice daily, with a 4-week continuous treatment cycle. Letrozole: 2.5 mg orally once daily, with a 4-week continuous treatment cycle.

Cohort 2 (dual-drug group) received: Apatinib: 250 mg orally once daily, with a 28-day treatment cycle. Letrozole: 2.5 mg orally once daily, with a 4-week continuous treatment cycle. reatment continued until disease progression, intolerable toxicity, or other protocol-specified reasons occurred.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* ECOG Performance Status score of 0 or 1;
* Epithelial ovarian cancer with platinum-sensitive recurrence (no restriction on histological type);
* Patients who have received first-line maintenance treatment with olaparib or niraparib (including but not limited to) and achieved complete response (CR) or partial response (PR) to second-line platinum-based chemotherapy;
* Availability of genetic testing results (BRCA1/2) and estrogen receptor (ER) testing results (ER positivity is defined as ≥ 1% of tumor cells staining positive for ER);
* Estimated survival of ≥ 6 months;
* Good function of major organs in the subject, with relevant test results meeting the following requirements within 7 days prior to enrollment:

Hematological tests (no blood transfusion or use of hematopoietic growth factors within 7 days prior to screening):

Hemoglobin (Hb) ≥ 90 g/L; Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L; Platelet count (PLT) ≥ 100×10⁹/L; White blood cell count (WBC) ≥ 3.0×10⁹/L and ≤ 15×10⁹/L;

Biochemical tests (no blood transfusion or albumin within 7 days prior to screening):

Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN); Alkaline phosphatase (ALP) ≤ 2.5 ULN; Total bilirubin (TBIL) ≤ 1.5 ULN; Serum creatinine (Cr) ≤ 1.5 ULN, with creatinine clearance (CrCL) ≥ 60 mL/min (Cockcroft-Gault formula); Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 ULN, with international normalized ratio (INR) ≤ 1.5 ULN (not receiving anticoagulant therapy); Urinalysis: Urine protein < 2+; if urine protein ≥ 2+, then 24-hour urine protein quantification must show protein ≤ 1 g; 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) for females < 470 ms;

* The subject voluntarily agrees to participate in this study, signs the informed consent form, and is willing to comply with the follow-up requirements.

Exclusion Criteria:

* Patients allergic to the trial drug or its excipients;
* Patients with active brain metastases;
* Patients who have received systemic treatment with traditional Chinese medicine or immunomodulatory agents (including thymosin, interferon, interleukin, excluding local use for pleural effusion control) within 2 weeks prior to the first dose;
* Patients with severe cardiovascular diseases: myocardial ischemia or myocardial infarction of grade II or above, uncontrolled arrhythmias (including QTc interval ≥ 470 ms); heart function of grade III-IV (according to the New York Heart Association [NYHA] classification), or echocardiogram showing left ventricular ejection fraction (LVEF) < 50%;
* Patients with severe infections within 4 weeks prior to the first dose (e.g., requiring intravenous antibiotics, antifungals, or antivirals), or unexplained fever > 38.5℃ during the screening period or prior to the first dose; or patients who have undergone major surgical procedures within 3 weeks prior to the first dose;
* Patients with type I diabetes mellitus whose blood glucose is controlled with insulin therapy may be eligible for this study;
* Patients undergoing systemic treatment with bronchodilators and having unsatisfactory asthma control are not eligible (patients with childhood asthma that has completely resolved and requires no intervention in adulthood may be included);
* Patients with human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis B, hepatitis C (positive hepatitis C antibody and HCV-RNA above the lower limit of detection of the assay), or co-infection with hepatitis B and C;
* Patients who have undergone or are planned to undergo solid organ or hematopoietic stem cell transplantation during the study period (excluding corneal transplantation);
* Patients currently participating in an interventional clinical study or who have received other investigational drugs or study devices within 4 weeks prior to the first dose; patients who have not fully recovered from toxicities and/or complications caused by any prior interventions (i.e., ≤ grade 1 or returned to baseline, excluding fatigue or alopecia);
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 110 mmHg despite optimal medical therapy);
* Coagulation abnormalities (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), tendency to bleed, or receiving thrombolytic or anticoagulant therapy;
* Urinalysis showing proteinuria ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;
* Patients with a history of allergy that may potentially cause hypersensitivity or intolerance to the trial drug or similar biologics;
* Patients with a history of substance abuse or psychiatric disorders that cannot be discontinued;
* Patients with a history of hereditary or acquired bleeding disorders or coagulopathies (eligibility to be determined by the investigator);
* Patients currently receiving strong CYP3A4 inhibitors (e.g., itraconazole, telithromycin, clarithromycin), moderate CYP3A4 inhibitors (e.g., ciprofloxacin, clarithromycin, fluconazole), strong CYP3A4 inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampin), or moderate CYP3A4 inducers (e.g., bosentan, modafinil). A washout period of 5 weeks is required for enzalutamide or phenobarbital, and 3 weeks for other drugs prior to the start of study treatment;
* Patients who have received small-molecule tyrosine kinase inhibitors (TKIs) for antiangiogenesis after achieving CR/PR with second-line platinum-based chemotherapy and using bevacizumab as maintenance therapy (patients previously treated with bevacizumab are allowed, but those treated with pazopanib, sorafenib, regorafenib, sunitinib, lenvatinib, anlotinib, etc., are not allowed);
* Patients with a history of cerebrovascular accident or transient ischemic attack within 6 months;
* Patients with other severe physical or psychiatric diseases or laboratory abnormalities that may increase the risk of participating in the study, interfere with study treatment or study results, or any other conditions deemed by the investigator as unsuitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival rate | 6 months
  The proportion of patients who survive without disease progression (defined as any increase in tumor size or death from any cause) within 6 months from the start of the formal treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 12 months
  Defined as the time from the start of formal treatment to the occurrence of disease progression (in any aspect) or death from any cause.
Overall Survival (OS) | 24 moths
  Defined as the time from the start of formal treatment to death from any cause, calculated in the intention-to-treat (ITT) population.
Time to First Subsequent Anti-Cancer Treatment (TFST) | 12 months
  The time from the start of formal treatment in the study to the initiation of the first subsequent anti-cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fengzhi Feng, PhD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No